CLINICAL TRIAL: NCT00264069
Title: Study ADH.E.R.E.: "Therapeutic ADHerence and Treatment Strategies: Mental Health Registry"
Brief Title: ADH.E.R.E.: Therapeutic ADHerence and Treatment Strategies: A Mental Health Registry
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Country Medical Director, Janssen-Cilag S.A., Spain
Other Study IDs: CR005755
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia; Bipolar Disorder; Depression; Personality Disorder
Keywords: Adherence; Compliance; Schizophrenia; Bipolar Disorder; Depression; Personality Disorders; Registry
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depression; Personality Disorders; Patient Compliance | interventions — Antipsychotic Agents; Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 001
  Interventions: Drug: antipsychotic
- 002
  Interventions: Drug: antidepressants

INTERVENTIONS:
Drug: antipsychotic — as prescribed
  Groups: 001
Drug: antidepressants — as prescribed
  Groups: 002

SUMMARY:
The purpose of this study is to find out how well new treatment plans are followed by outpatients with major mental illnesses (schizophrenia, bipolar disorder, depression, personality disorder) and to determine the relationship between a diagnosis of schizophrenia and compliance with a treatment plan.

DETAILED DESCRIPTION:
Compliance (which refers to how well one follows a prescribed medication or therapy) varies among all types of diseases, but it is generally low for those outpatients with major mental illness. This leads to relapses and worsening of their condition, and worsening of their condition may lead to poor compliance. The purpose of the study is to record, analyze, and report how well patients with major mental illness in an outpatient setting follow the prescribed treatment plan for the first few months of a new treatment strategy (either a first-time therapy plan or a change to a therapy plan). Therapy plans include psychiatric counseling (psychotherapy), visits to the outpatient clinic, and taking prescribed drugs. "Compliance" is defined as actually doing what the plan says, including attending therapy sessions, going for clinic visits, and taking necessary medication. The study will look for individual factors for each patient that might influence lack of compliance, and then see whether some of the individual factors predict a lack of compliance in the group as a whole, which includes approximately 2500 patients. These factors include a diagnosis of schizophrenia compared with a diagnosis of another major mental illness such as depression, bipolar disorder, or personality disorder. Social and personal factors will also be recorded and analyzed to see whether they influence the patient's ability to follow the treatment plan. Examples are age, sex, education, race, urban versus rural lifestyle, family supportiveness, and substance abuse status. Other factors to be studied that may vary between patients who are either good, average, or poor at following their treatment plan include the number of hospital admissions for each patient, how long it has been since their last hospitalization, and the reason why their new therapy plan was changed or started. The study will also try to determine how physicians confirm the patient's reports of their adherence to their treatment plan. A physician may take blood to measure levels of the drug, count a patient's pills or injections, or simply ask the patient or a family member. Researchers will compare compliance when different classes of drugs are prescribed, such as antidepressants and antipsychotics, to determine whether a particular group of drugs is associated with improved compliance. The safety and effectiveness of the drugs prescribed might also influence whether patients take their medication, so these factors will be evaluated. Adverse events (unintended and undesirable effects that might be due to the treatments) will be recorded for each patient over the 3 months of the study, and the physician will record the results of a Global Clinical Impression scale that ranges from "No Illness" to "Extreme Illness" to record an overall impression of the patient's illness before and after treatment. Antipsychotics and antidepressants, as used in routine clinical practice. Study duration is 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients diagnosed with schizophrenia, bipolar disorder or depression according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) classification characteristics who have been given a new therapy plan (that may include drug treatment for mental illness, visits to a mental health care worker, or other treatments such as non-medication type of treatments)
* Patients either scheduled for treatment in the next 3 months or already treated for the past 3 months

Exclusion Criteria:

* Patients with psychiatry pathology other than Schizophrenia or schizoaffective disorder/ bipolar disease/major depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients diagnosed with schizophrenia, bipolar disorder or depression according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) classification characteristics who have been given a new therapy plan (that may include drug treatment for mental illness, visits to a mental health care worker, or other treatments such as non-medication type of treatments); patients either scheduled for treatment in the next 3 months or already treated for the past 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 2622 (Actual)
Dates: Start 2005-06; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Comparison of compliance with different classes of drugs (such as antidepressants and antipsychotics), to determine whether a particular group of drugs is associated with improved compliance. | 3 months

SECONDARY OUTCOMES:
Comparison of compliance with different classes of drugs (such as antidepressants and antipsychotics), to determine whether a particular group of drugs is associated with improved compliance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.

REFERENCES:
- See also: Treatment Adherence and Strategies: A Mental Illness Registry (ADHERE study) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=280&filename=CR005755_CSR.pdf